CLINICAL TRIAL: NCT00681733
Title: A Study Of Metabolic Factors And Efficacy Of Pentoxifylline Versus Pioglitazone In Lean And Obese Nash (Non-Alcoholic Steatohepatitis) Patients.
Brief Title: Pentoxifylline Versus Pioglitazone In Non-Alcoholic Steatohepatiti (NASH)
Acronym: NASH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Govind Ballabh Pant Hospital (Other Government)
Responsible Party: Dr. B C Sharma, professor, G B Pant Hospital, New Delhi, G B Pant Hospital, New Delhi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: drakchaudhary; drakchaudhary
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Last update posted 2008-05-21 (Estimated); Status verified 2008-05

CONDITIONS: Metabolic Parameters and Liver Histology
Keywords: NASH Pentoxifylline Pioglitazone
MeSH Terms: interventions — Pioglitazone; Pentoxifylline

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Pioglitazone
  Interventions: Drug: Pioglitazone
- B (Active Comparator): Pentoxifylline
  Interventions: Drug: Pentoxifylline

INTERVENTIONS:
Drug: Pioglitazone — Pentoxifylline 1200mg/day in 3 divided doses. Pioglitazone 30 mg/day in single dose
  Other Names: Pentoxifylline - Trental; Pioglitazone - Piosys, Pioglar
  Arms: A
Drug: Pioglitazone — 30 mg OD
  Other Names: Pioglar
  Arms: A
Drug: Pentoxifylline — 1200 mg/d
  Other Names: Trental
  Arms: B

SUMMARY:
1. To assess the metabolic factors in lean and obese patients with NASH.
2. To compare the efficacy of pentoxifylline versus pioglitazone on the metabolic profile and liver histology of NASH patients.

DETAILED DESCRIPTION:
A total of 40 patients with biopsy proven NASH will be enrolled.

Inclusion criteria

* Abdominal USG showing diffusely echogenic liver suggestive of fatty infiltration of liver.
* ALT > 1.2 times the upper limit of normal for > 6 months.(atleast three readings one month apart)
* Liver Biopsy showing steatosis affecting >10% of hepatocytes with necroinflammatory activity, ballooning hepatocytes &/ or fibrosis.

Exclusion criteria

* Alcohol intake of more than 20g/wk
* Evidence of viral/ autoimmune hepatitis
* PBC (Primary biliary cirrhosis)
* Biliary obstrution
* Wilson disease
* Haemchromatosis
* Decompensated cirrhosis
* Drug ingestion of the follwing drugs for a period of more than 4 weeks during past 6 weeks

  * Amiodarone
  * Methotrexate
  * Perhexiline
  * Glucocorticoids
  * Estrogens
  * Tamoxifen
  * Nifedipine
  * Diltiazem
  * Tamoxifen
* DM Type I

STUDY DESIGN

The study will be divided into two parts Part A and Part B.

Part A

* A cross-sectional study of metabolic profile will be done at the enrollment with a detailed physical examination and laboratory investigations and certain specific tests for non-alcoholic steatohepatitis.
* At enrollment following characteristics will be included-
* Prior history of Diabetes, Hypertension, Dyslipidemia, Coronary artery disease.
* Age, sex, weight, height, BMI(body mass index), waist & hip circumference.
* USG abdomen
* LFT
* Fasting glucose, post-prandial blood sugar/oral GTT(glucose tolerance test)
* Fasting insulin level
* Fasting C- peptide
* HOMA-IR (Homeostasis Model Assessment-insulin resistance)
* Fasting lipid profile
* Fasting TNF- α
* Fasting Adiponectin
* Fasting Leptin
* Liver biopsy
* Waist will be measured with soft tape on standing subjects midway between the lowest rib and iliac spine.
* BMI of every patient will be calculated.
* Lean patient will be defined as BMI of 18.5- 22.9 kg/m2
* Overweight as ≥ 23- 24.9 kg/m2
* Obese as ≥ 25 kg/m2
* Lean patient will be further categorized as

  1. Normal waist circumference (< 90cm for men, < 80 cm for women)
  2. Abnormal waist circumference (more than the above mentioned criteria)
* Insulin resistance will be calculated by HOMA-IR

  * Fasting serum insulin (μIU/ ml) x Fasting serum glucose(mmol/l) ÷ 22.5 HOMA-IR >2 will be taken as insulin resistance.
* TNF- α, adiponectin and leptin will be measured by ELISA method using standard kits.
* Liver biopsy will be analyzed by pathologist at the time of enrollment into the study. Histology reporting will be done by the method given by Brunt et al.23

Part B.

A Prospective Randomized Controlled Trial comparing efficacy of Pentoxyphylline versus Pioglitazone will be done.

A total of 40 NASH patients (lean and obese) will be enrolled. All will be advised dietary and exercise protocol. Twenty patients will be randomized to receive Pentoxifylline in a dose of 1200mg/day in 3 divided doses. Another twenty patients will receive Pioglitazone in a dose of 30 mg/day. The subjects will be randomly assigned to receive either pentoxifylline or pioglitazone (randomization will be computer-generated). Patients will be followed with liver biochemistry at monthly interval for initial 3 months and subsequently at 3 month interval. .Liver biopsy will be repeated at the end of 6 months of therapy. The pathologist will blinded to the drug administered to the NASH patients.

Adverse events associated with Pentoxifylline and pioglitazone will be inquired and recorded on follow-up visits. The known side-effects of Pentoxiphylline are nausea, headache, vomiting, dyspepsia, bloating, flushing, vertigo and gastroesophageal reflux and that of Pioglitazone are myalgia, weight gain and pedal edema.

END POINT OF THE STUDY

1. Repeat metabolic parameters and liver biopsy will be done at the end of 6 months.
2. Improvement by 50% or normalization of aminotransferase at the end of the study will be compared to the baseline.
3. Histology will be compared with the repeat liver biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy proven NASH will be enrolled. Abdominal USG showing diffusely echogenic liver suggestive of fatty infiltration of liver.
* ALT > 1.2 times the upper limit of normal for > 6 months.(atleast three readings one month apart)
* Liver Biopsy showing steatosis affecting >10% of hepatocytes with necroinflammatory activity, ballooning hepatocytes &/ or fibrosis.

Exclusion Criteria:

* Alcohol intake of more than 20g/wk
* Evidence of viral/ autoimmune hepatitis
* PBC (Primary biliary cirrhosis)
* Biliary obstrution
* Wilson disease
* Haemchromatosis
* Decompensated cirrhosis
* Drug ingestion of the follwing drugs for a period of more than 4 weeks during past 6 weeks - Amiodarone, Methotrexate, Perhexiline, Glucocorticoids, Estrogens, Tamoxifen, Nifedipine, Diltiazem, Tamoxifen.
* DM Type I

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in metabolic profile and histology | 6 months

SECONDARY OUTCOMES:
Side effects | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Barjesh Ch Sharma, MD, DM, Principal Investigator — G B Pant Hospital Hospital, New Delhi
Locations (1):
- Dr. Barjesh Chander Sharma, New Delhi, New Delhi, India